CLINICAL TRIAL: NCT05334394
Title: The Effect of Mulligan Mobilization Technique on Balance, Pain and Functionality in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Kubra Bali, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2868
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Chronic Low-back Pain; Lumbal Disc Herniation; Imbalance
Keywords: Balance; Chronic Low Back Pain; Exercise; Lumbal Disc Herniation; Manual Therapy; Mulligan Mobilization
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Group (Experimental)
  Interventions: Other: Mulligan Technique
- Control Group (Experimental)
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Mulligan Technique — Mulligan suggested that injuries or sprains can cause a minor positional error in a joint, thereby causing limitations in physiological movement. Unique to this concept is mobilization of the spine while weight bearing and directing the mobilization parallel to the spinal facet planes. Although it includes various mobilization techniques, one of the most important techniques, motion co-mobilization, is the SNAG's technique, which includes the application of accessory passive gliding to the lumbar vertebra while the patient performs active movement simultaneously.
  Arms: Mulligan Group
Other: Exercise Therapy — Exercise is recommended by physical therapists for most chronic low back pain patients.
  Arms: Control Group

SUMMARY:
This study was aimed to investigate the effectiveness of mulligan mobilization technique on balance, pain and functionality in patients with chronic low back pain and to compare it with exercise.37 patients aged between 18-65 who applied to Fındıkzade Medipol Hospital were included in the study. The individuals participating in the study were divided into two groups, 18 control and 19 mulligan groups, according to the randomization table. The intervention was performed 3 times a week for 4 weeks. Conventional physiotherapy and exercise program accompanied by a physiotherapist were applied to the control group, and conventional physiotherapy and mulligan mobilization technique were applied to the mulligan group. Conventional physiotherapy methods included ultrasound (US), Transcutaneous Electrical Nerve Stimulation (TENS), and hotpack. The patients were evaluated with TecnoBody Static Balance Device, algometer, electrogoniometer, visual analog scale, Oswestry Low Back Pain Disability Questionnaire before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing non-specific chronic low back pain for more than 3 months
* The diagnosis has been confirmed by the Health Board Report
* Be over 18 years old
* Be younger than 65 years old
* Pain of at least 2 severity according to VAS
* Voluntarily agree to participate in the study

Exclusion Criteria:

* Previous lumbar trauma or operation
* Long-term use of corticosteroids
* Cancer
* Pregnancy
* Osteoporosis
* Systemic Diseases
* Spinal Deformities
* Lumbal Stenosis
* Ankylozone Spondylitis
* Spondylolisthesis
* Spinal Deformities
* Lumbal Stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
TecnoBody Static Balance Device Measurements | 5 Minutes
  TecnoBody Stability Easy is a stabilometric system consisting of three highly sensitive sensors. The system is based on continuous observation of the foot pressure center (COP). By recording the postural oscillations of the body as a function of time, detailed information about the postural system is obtained
Pressure Pain-Threshold Measurements with Algometer | 5 Minutes
  It is a device used to evaluate the sensitivity to pain and to determine the perception of pressure. The pressure algometer has proven useful in evaluating fibrositis and hypersensitive spots, trigger points, arthritis activation, and visceral pain-pressure sensitivity.
Electrogoniometer | 5 Minutes
  It is an evaluation tool used to record the objective measurement of joint range of motion.

SECONDARY OUTCOMES:
Visual Analog Scale | 1 Minutes
  Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically into digital. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his / her condition is appropriate by drawing a line or by placing a dot or marking.
Oswestry Disability Index | 10 Minutes
  The Oswestry Disability Index is a commonly used outcome measure to detect perceived disability in patients with low back pain. It consists of 10 questions, each of which is scored between 0 and 5, assessing the degree of pain, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and change in pain. The minimum score obtained from the scale is 0, and the maximum score is 50. 0-4 points as no disability, 5-14 points as mild, 15-24 points as moderate, 25-34 points as severe and 35-50 points as complete functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Bali, Licenced, Principal Investigator — Medipol University
Locations (1):
- Fındıkzade Medipol Hospital, Istanbul, Fındıkzade, Turkey (Türkiye)